CLINICAL TRIAL: NCT03418194
Title: Effects of Transcutaneous Acupoint Electrical Stimulation on Postoperative Heart Rate Variability and High-sensitive Cardiac Troponin of Elderly Patients With Coronary Heart Disease
Brief Title: Effects of Transcutaneous Acupoint Electrical Stimulation on Postoperative HRV and Hs-cTnT of Elderly With CHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebei Medical University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAESOFLHZ
Record Dates: First submitted 2018-01-25; First posted 2018-02-01 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Coronary Artery Disease; Anesthesia
Keywords: Anesthesia, General
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAES group (Experimental): Patients in group TAES group received transcutaneous acupoint electrical stimulation (disperse-dense waves, frequency 4/20Hz) at the points of PC6 (Neiguan) and PC4 (Ximen) from 30 min before anesthesia induction to the end of surgery,
  Interventions: Procedure: transcutaneous acupoint electrical stimulation
- control group (Placebo Comparator): Patients in group C received electrode plate atthe points of PC6 (Neiguan) and PC4 (Ximen) without any electrical stimulation.
  Interventions: Procedure: sham transcutaneous acupoint electrical stimulation

INTERVENTIONS:
Procedure: transcutaneous acupoint electrical stimulation — Transcutaneous acupoint electrical stimulation(TAES) is a kind of noninvasive therapy similar to acupuncture and moxibustion. Its physiological effect is similar to that of electroacupuncture and hand acupuncture which is a Chinese traditonal therapy using acupuncture.
  Arms: TAES group
Procedure: sham transcutaneous acupoint electrical stimulation — Sham transcutaneous acupoint electrical stimulation is the same procedure as transcutaneous acupoint electrical stimulation at points without electronic stimulation.
  Arms: control group

SUMMARY:
The aim of this study was to observe the effect of transcutaneous acupoint electrical stimulation (TAES) on postoperative heart rate variability and high-sensitive cardiac troponin T of elderly patients with coronary heart disease.

DETAILED DESCRIPTION:
General anesthesia can inhibit sympathetic nerve activity and attenuate stress response, but it also inhibits vagus nerve activity. The decrease of vagus nerve activity can cause cardiovascular complications, especially ventricular arrhythmia in patients with coronary heart disease. Some study have shown that electrical stimulation of transcutaneous acupoints can regulate the function of autonomic nervous system and enhance the activity of vagus nerve so as to protect myocardial tissue. But the effect on autonomic nervous function and myocardial injury markers in elderly patients with coronary heart disease was not reported. Heart rate variability (HRV) is a noninvasive and reliable index reflecting cardiac autonomic nervous function. High-sensitive cardiac troponin hs-cTnT is the best myocardial injury marker.

The investigators plan to recruite 150 patients with coronary heart disease of both sexes, aged 65-80 yr, undergoing elective lumbar decompression and fusion internal fixation surgery. They will be randomly divided into 2 groups(n=75 each)using random number table : control group ( group C ) and TAES group (group T). Patients in group T receive TEAS (disperse-dense waves, frequency 4/20Hz) at the points of PC6 (Neiguan) and PC4 (Ximen) from 30 min before anesthesia induction to the end of surgery, the optimal intensity will be adjusted to maintain a slight twitching of the midfinger or ring finger (De-Qi response). Patients in group C receive electrode plate at the same acupoints without any electrical stimulation. Heart rate variability will be collected on 1 day before surgery, 1, 3 and 5d after surgery. 3mL of venous blood will be collected before the induction of anesthesia, 1, 3 and 5d after surgery, the serum will be isolated for the measurement of serum concentration of high-sensitive troponin T (hs-cTnT)、CK、CRP.

ELIGIBILITY:
Inclusion Criteria:

* Stable angina pectoris
* Slilent myocardial ischemia
* Remote myocardial infarction

Exclusion Criteria:

* Congenital heart disease
* Have a history of cardiac surgery
* Frequent ventricular / atrial premature beats, atrial fibrillation and other serious arrhythmia
* Heart conduction diseases
* Antiarrhythmic drugs used
* Temporary and permanent pacemaker used
* Intraoperative blood loss>800ml

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 137 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
High-sensitive cardiac troponin T | 1 week
  Cardiac troponin T are components of the contractile apparatus of myocardial cells and are expressed almost exclusively in the heart. High-sensitive cardiac troponin T is cardiac troponin T mesured by high-sensitive method.

SECONDARY OUTCOMES:
heart rate variability | 1 week
  Heart rate variability (HRV) has been verified as a noninvasive indicator of the autonomic nervous system.
CK | 1 week
  CK is an indicator that reflects the amplitude of operation injury in spine surgery. 1, 3 and 5d after surgery, the serum concentration of CK.
CRP | 1 week
  CRP is a non-specific biomarker of inflammation which has been described as a risk factor for cardiovascular disease. 1, 3 and 5d after surgery, the serum concentration of CRP.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Wang, MD, PhD, Study Chair — Third Hospital of Hebei Medical Universit Department of Anesthesiology; Huizhou li, M.D, Study Director — Third Hospital of Hebei Medical Universit Department of Anesthesiology; Chuan Wu, M.D, Principal Investigator — Third Hospital of Hebei Medical Universit Department of Anesthesiology
Locations (1):
- Third Hospital of Hebei Medical Universit, Shijiazhuang, Hebei, China

REFERENCES:
- [Result] Mazzeo AT, La Monaca E, Di Leo R, Vita G, Santamaria LB. Heart rate variability: a diagnostic and prognostic tool in anesthesia and intensive care. Acta Anaesthesiol Scand. 2011 Aug;55(7):797-811. doi: 10.1111/j.1399-6576.2011.02466.x. Epub 2011 Jun 9. PMID 21658013
- [Result] Writing Committee for the VISION Study Investigators; Devereaux PJ, Biccard BM, Sigamani A, Xavier D, Chan MTV, Srinathan SK, Walsh M, Abraham V, Pearse R, Wang CY, Sessler DI, Kurz A, Szczeklik W, Berwanger O, Villar JC, Malaga G, Garg AX, Chow CK, Ackland G, Patel A, Borges FK, Belley-Cote EP, Duceppe E, Spence J, Tandon V, Williams C, Sapsford RJ, Polanczyk CA, Tiboni M, Alonso-Coello P, Faruqui A, Heels-Ansdell D, Lamy A, Whitlock R, LeManach Y, Roshanov PS, McGillion M, Kavsak P, McQueen MJ, Thabane L, Rodseth RN, Buse GAL, Bhandari M, Garutti I, Jacka MJ, Schunemann HJ, Cortes OL, Coriat P, Dvirnik N, Botto F, Pettit S, Jaffe AS, Guyatt GH. Association of Postoperative High-Sensitivity Troponin Levels With Myocardial Injury and 30-Day Mortality Among Patients Undergoing Noncardiac Surgery. JAMA. 2017 Apr 25;317(16):1642-1651. doi: 10.1001/jama.2017.4360. PMID 28444280